CLINICAL TRIAL: NCT03409679
Title: A Multicenter, Open-label, Randomized, Active-controlled, Parallel Group, Pivotal Study to Investigate the Efficacy, Safety and Tolerability, and Pharmacokinetics of Murepavadin Combined With One Anti-pseudomonal Antibiotic Versus Two Anti-pseudomonal Antibiotics in Adult Subjects With Ventilator-associated Bacterial Pneumonia Suspected or Confirmed to be Due to Pseudomonas Aeruginosa
Brief Title: Pivotal Study in VAP Suspected or Confirmed to be Due to Pseudomonas Aeruginosa
Acronym: PRISM-MDR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety data review
Sponsor: Polyphor Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POL7080-011
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-05

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — murepavadin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Murepavadin (Experimental): Murepavadin IV + one anti-pseudomonal antibiotic
  Interventions: Drug: Murepavadin
- Two anti-pseudomonal antibiotics (Active Comparator): Association of 2 anti-pseudomonal antibiotics
  Interventions: Drug: Two anti-pseudomonal antibiotics

INTERVENTIONS:
Drug: Murepavadin — Murepavadin IV every 8 hours + 1 anti-pseudomonal antibiotic (Piperacillin-tazobactam, ceftazidine, cefepime, meropenem, amikacin, ciprofoxacin, levofloxacin, colistin)
  Arms: Murepavadin
Drug: Two anti-pseudomonal antibiotics — Piperacillin-tazobactam, ceftazidine, cefepime, meropenem, amikacin, ciprofoxacin, levofloxacin, colistin
  Arms: Two anti-pseudomonal antibiotics

SUMMARY:
This is a phase 3, multicenter, open-label, randomized active-controlled, parallel group to investigate the efficacy, safety and tolerability, and pharmacokinetics of intravenous murepavadin combined with of one anti-pseudononas antibiotic with that of two anti-pseudomonas antibiotics in the treatment of ventilator-associated bacterial pneumonia (VABP) in adult subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has received mechanical ventilation for at least 48h at the time of the randomisation
* Acute Physiology and Chronic Health Evaluation (APACHE) of 8 to 30, inclusive, within 24h prior to randomization
* Presence of new or progressive infiltrate on chest X-ray
* Presence of clinical criteria consistent with VABP
* High probability of VABP caused by Pseudomonas aeriginosa

Key Exclusion Criteria:

* Known or suspected community-acquired bacterial pneumonia or viral, fungal, or parasitic pneumonia
* Known hypersensitivity or contra-indications to beta-lactam antibiotics, aminoglycosides, quinolones, colistin, or subjects with a clinically significant history of anaphylactic reaction
* Severe liver or renal impairment
* Women who are pregnant or nursing, or who are of chilbearing potential and unwilling to use acceptable method of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate | 21-24 days after start of study treatment

CONTACTS AND LOCATIONS:
Locations (61):
- United States (3):
  - Research site, Chicago, Illinois
  - Research site, Springfield, Missouri
  - Research site, Greensboro, North Carolina
- Brazil (5):
  - Research Site 1, Belo Horizonte
  - Research Site 2, Belo Horizonte
  - Research Site, Itaquaquecetuba
  - Research Site, Porto Alegre
  - Research Site, São José do Rio Preto
- Croatia (2):
  - Research site 1, Zagreb
  - Research site 2, Zagreb
- Estonia (3):
  - Research site, Tallinn
  - Reasearch site, Tartu
  - Reasearch site, Võru
- France (8):
  - Research site, Lille
  - Reasearch site, Limoges
  - Research site, Lyon
  - Reasearch site, Nice
  - Research site 1, Paris
  - Research site 2, Paris
  - Research site 3, Paris
  - Research site, Pierre-Bénite
- Greece (6):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site 1, Larissa
  - Research Site 2, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hungary (6):
  - Reasearch site, Budapest, BU
  - Research site, Budapest, BU
  - Reasearch site, Ózd, BZ
  - Research Site, Kistarcsa
  - Research Site, Székesfehérvár
  - Research Site, Vác
- Israel (6):
  - Research site, Jerusalem, JM
  - Research site, Nahariya, Z
  - Research site, Tiberias, Z
  - Research site, Petah Tikva
  - Research site, Safed
  - Research site, Tel Litwinsky
- Mexico (3):
  - Research Site 1, Guadalajara
  - Research Site 2, Guadalajara
  - Research Site, Monterrey
- South Africa (4):
  - Research site 1, Pretoria, Gauteng
  - Research Site, Cape Town
  - Research Site 2, Pretoria
  - Research Site, Pretoria
- South Korea (8):
  - Research Site, Ansansi Danweongu
  - Research Site, Gangwon-do
  - Research site, Gyeongsang
  - Research site, Incheon
  - Research site 1, Seoul
  - Research site 2, Seoul
  - Research Site 3, Seoul
  - Research site, Seoul
- Spain (3):
  - Research site, Barcelona, B
  - Research site, Terrassa, B
  - Research site, Girona
- Thailand (4):
  - Research Site 1, Bangkok
  - Research Site 2, Bangkok
  - Research Site, Khon Kaen
  - Research Site, Nonthaburi